CLINICAL TRIAL: NCT04841083
Title: A Real World Evaluation of the Allay Lamp in Reducing Headache Symptoms and Frequency
Brief Title: Narrow Band Green Light and Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedanta Research (Other)
Responsible Party: Principal Investigator, Michael Reed, Managing Director, Vedanta Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL-20-01
Record Dates: First submitted 2021-04-01; First posted 2021-04-12 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allay lamp (narrow band green light) (Experimental): Subjects who purchased the Allay Lamp are asked to document the effects of spending time in the narrow band of green light it emits, on their headache or any of its associated symptoms.
  Interventions: Device: Allay Lamp

INTERVENTIONS:
Device: Allay Lamp — The Allay Lamp is a consumer product currently available and widely used in the US. It emits low intensity (1-10 lux) narrow band (20 nm) green light (peak wavelength 520 nm) that is marketed as non-irritating to users. In that context, it is not a medical device and does not require a 510(k).

SUMMARY:
Study volunteers are asked to use the Allay Lamp routinely during the 6-week study period. A web based survey is provided when the Lamp is purchased for study volunteers to complete. A daily usage paper diary is sent with the lamp so that volunteers can keep track of the frequency and duration of lamp usage and any noticeable benefits. At the end of six weeks a second survey is sent to study volunteers to capture their perceptions of potential lamp benefits with respect to headache frequency and their experience of migraine specific symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults with headaches or migraines.

Exclusion Criteria:

* Not having headaches or migraines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Change in number of headache days per week | Change from baseline at 6 weeks
  Number of days with headache per week without and with using the Allay lamp
Change in number of headache days per month | Changes from baseline at weeks 3-6 of using the Allay lamp
  Number of days with headache per month without and with using the Allay lamp
Change in frequency of experiencing photophobia | Changes from baseline at 6 weeks of using the Allay Lamp.
  Assessing frequency of photophobia during days with headache as depicted by participants using the following options: (1)never, rarely, (2)less than half, (3)half or more, (4)nearly all the time.
Change in headache severity | Changes from baseline at 6 weeks of using the Allay lamp
  Assessing headache severity while using the Allay lamp. Improvement is determined by the number of times participants answer Yes or NO in their daily diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Vendata Research, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Lipton RB, Melo-Carrillo A, Severs M, Reed M, Ashina S, Houle T, Burstein R. Narrow band green light effects on headache, photophobia, sleep, and anxiety among migraine patients: an open-label study conducted online using daily headache diary. Front Neurol. 2023 Oct 4;14:1282236. doi: 10.3389/fneur.2023.1282236. eCollection 2023. PMID 37859647